CLINICAL TRIAL: NCT05046275
Title: The "Motoric Cognitive Risk" Syndrome in the Quebec Population: Results From the NuAge Study - Sub-study: The Biological Underpinnings of Motoric Cognitive Risk Syndrome: a Multicenter Study
Brief Title: MCR Syndrome in Quebec : Results From NuAge Study
Status: Active, not recruiting | Type: Observational
Sponsor: Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal (Other Government)
Responsible Party: Principal Investigator, Olivier Beauchet, MD, PhD, Senior researcher, Director of laboratory, Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal
Other Study IDs: 2021-245
Record Dates: First submitted 2021-09-08; First posted 2021-09-16 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Motoric Cognitive Risk Syndrome; Aging Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MCR syndroms: Summarize of participants' characteristics using means and standard deviations or frequencies and percentages First, prevalence of MCR syndrome will be determined by classifying participants into MCR and non-MCR syndrome groups. Second, between-group comparisons of participants' characteristics will be performed using unpaired t-test, Mann-Whitney, analysis of variance with LSD correction or Chi-square test, as appropriate. Third, multiple regressions will be performed to examine the association between MCR syndrome (dependent variable) and cardio-vascular risk factors and/or diseases (independent variables) adjusted on participants' characteristics. Fourth, the incidence of MCR syndrome during the follow-up period of NuAge study will be reported. Fifth, regression will be performed to examine the association between MCR syndrome (dependent variable) and cognitive decline as well cognitive impairment (independent variables, separated model) adjusted on participants' characteristics.
  Interventions: Other: Data analysis
- Non MCR syndroms: Summarize of participants' characteristics using means and standard deviations or frequencies and percentages First, prevalence of MCR syndrome will be determined by classifying participants into MCR and non-MCR syndrome groups. Second, between-group comparisons of participants' characteristics will be performed using unpaired t-test, Mann-Whitney, analysis of variance with LSD correction or Chi-square test, as appropriate. Third, multiple regressions will be performed to examine the association between MCR syndrome (dependent variable) and cardio-vascular risk factors and/or diseases (independent variables) adjusted on participants' characteristics. Fourth, the incidence of MCR syndrome during the follow-up period of NuAge study will be reported. Fifth, regression will be performed to examine the association between MCR syndrome (dependent variable) and cognitive decline as well cognitive impairment (independent variables, separated model) adjusted on participants' characteristics.
  Interventions: Other: Data analysis

INTERVENTIONS:
Other: Data analysis — No intervention, data analysis only

SUMMARY:
The overall objective of the proposal is to examine the epidemiology of the newly reported "motoric cognitive risk" (MCR) syndrome, which is a pre-dementia syndrome combining subjective cognitive complaint (i.e.; memory complaint) with objective slow gait speed, in the Quebec elderly population.

Cognition and locomotion are two human abilities controlled by the brain. Their decline is highly prevalent with physiological and pathological aging, and is greater than the simple sum of their respective prevalence, suggesting a complex age-related interplay between cognition and locomotion. Both declines in cognition and locomotion are associated, furthermore the temporal nature of their association has been unclear for a long time. Recently, a systematic review and meta-analysis has provided evidence that poor gait performance predicts dementia and, in particular, has demonstrated that MCR syndrome is a pre-dementia syndrome, suggesting that low gait performance is the first symptom of dementia. The uniqueness of MCR syndrome is that it does not rely on a complex evaluation or laboratory investigations. Indeed, this syndrome combined subjective cognitive complaint and objective slow gait speed, and is easy to apply in population-based settings.

Prevalence and incidence of MCR syndrome, as well as its association with incidence of cognitive decline and impairment, have never been reported in Canada. Nutrition as a determinant of successful aging: The Quebec longitudinal Study (the NuAge study) is a Quebec population-based observational cohort study performed in healthy older community-dwellers adults which provides a unique opportunity to: 1) obtain reliable estimates of MCR syndrome prevalence and incidence, 2) determine the distribution of clinical and biological (blood biomarkers and genetic) characteristics associated with MCR syndrome, 3) examine the association of MCR syndrome and its biological characteristics with cognitive decline and incidence of cognitive impairment in the Quebec elderly population.

ELIGIBILITY:
Inclusion Criteria:

* All included participants of NuAge Study

Exclusion Criteria:

* no information about cognitive complaint in NuAge database
* no measure of walking speed in NuAge database
* no follow-up completed in NuAge database

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: All included participants of NuAge Study were healthy and, in particular, they were cognitively intact at baseline and had no mobility disability.
Sampling Method: Non-Probability Sample
Enrollment: 1741 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2025-11-02 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
prevalence of MCR syndrome | 3 years
  Diagnosis of MCR syndrome following Verghese et al. criteria

SECONDARY OUTCOMES:
Cognitive decline and impairment | 3 years
  Modified Mini-Mental State (3MS) in the NuAge study.
Covariates | 3 years
  Cardio-vascular risk factors and diseases assessed using reported health condition
Covariates | 3 years
  Cardio-vascular risk factors and diseases assessed using physical examination: body mass index
Covariates | 3 years
  Cardio-vascular risk factors and diseases assessed using physical examination: hip waist ratio from hip and waist circumference
Covariates | 3 years
  Cardio-vascular risk factors and diseases assessed using physical examination: blood pressure (value of systolic, diastolic when participants are seated in an upright position in a chair)
Biological characteristics | 3 years
  we selected biomarkers that consistently show associations with clinical risk factors for MCR : IL-6, high-sensitivity CRP and Malondialdehyde (MDA). These biomarkers are associated with individual MCR components. CRP was associated with plaques. Inflammation is hypothesized to be a precursor to neurofibrillary tangles and amyloid plaques; hallmarks of AD. Oxidative stress damage is elevated in vulnerable brain regions in early AD and MCI.
  We propose a multi-level examination of vascular pathways in MCR including biomarkers (CRP and homocysteine).
  We include homocysteine, a vascular biomarker, linked to gait and cognitive deficits in other studies.
Genetic approach | 3 years
  we propose to derive polygenic risk scores for cognitive and obesity phenotypes in NuAge, and to examine its predictive validity for MCR syndrome and incident cognitive impairment

CONTACTS AND LOCATIONS:
Locations (1):
- CRIUGM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No